CLINICAL TRIAL: NCT02828189
Title: Efficacy of Therapeutic Exercise in Modulating Cancer-Related Fatigue in Women After Breast Cancer Treatment
Brief Title: Therapeutic Exercise in Cancer-Related Fatigue in Women After Breast Cancer Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Virginia Prieto Gómez, Teacher care and research in physiotherapy Unit. Department of Physiotherapy. University of Alcala., University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FPSM_UAH_VPG_2
Record Dates: First submitted 2016-06-29; First posted 2016-07-11 (Estimated); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Fatigue; Breast Cancer
Keywords: Physical Therapy Modalities; Breast Cancer Treatment; Exercise Therapy; Dyspnea
MeSH Terms: conditions — Fatigue; Breast Neoplasms; Dyspnea | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical Exercise (Active Comparator): The protocol consists in:
  * Physical Exercise according to their preferences.
  * Therapeutic Education related to Health Habits and Physical Exercise.
  Interventions: Other: Physical Exercise; Behavioral: Therapeutic Education
- Therapeutic Exercise-Physiotherapy (Experimental): The protocol consists in:
  * Cardiovascular exercise.
  * Force-Resistance Exercises of the principals muscle groups of the lower limbs, upper limbs and trunk.
  * Muscle Stretches.
  * Therapeutic Education related to Health Habits and Physical Exercise.
  Interventions: Behavioral: Therapeutic Education; Other: Therapeutic exercise-Physiotherapy

INTERVENTIONS:
Other: Physical Exercise — The patients were instructed to perform autonomous physical exercise program based preferences (progressive march on flat ground, dancing, cycling, etc.). They will receive written information. The program is 9 weeks with a frequency of 3 days per week and sessions about 50 minutes long.
  Other Names: Exercise
  Arms: Physical Exercise
Behavioral: Therapeutic Education — Individual Therapeutic Education about healthy habits and exercise on breast cancer.
  Other Names: Hygienic and behavioral advises
Other: Therapeutic exercise-Physiotherapy — 1. Cardiovascular exercise
  2. Individualized progressive strength and resistance exercises of principals muscle groups of the lower limbs, upper limbs and trunk.
  3. Flexibilization exercises
  Other Names: Physiotherapy exercise
  Arms: Therapeutic Exercise-Physiotherapy

SUMMARY:
The main objective of this study is to determine whether the proposed program of therapeutic exercise is effective in improving fatigue, more than the exercise unsupervised depending on their preferences, in women treated for breast cancer.

DETAILED DESCRIPTION:
Introduction: The prevalence of cancer-related fatigue in women treated for breast cancer is about 30% having significant effects in reducing their quality of life. There is evidence of the presence of sleep problems and immune response. Several studies claim that physical exercise is effective during and after treatment of the disease as it improves the quality of life, cardiorespiratory function, physical functioning and symptoms of fatigue although not always found significant differences between intervention groups exercises compared with a control group. Although the results of these studies are promising, generally present methodological biases as small sample size, absence of masking, heterogeneous groups, lack of monitoring short and long term and especially lack of specificity in relation to prescribed exercise ( frequency, intensity, time and type of exercise).

Subjects and methods: A randomized clinical trial, the examiner being blinded unaware of the intervention group to which subjects were assigned. Participants will be randomly assigned to two groups:

An experimental group, where the participants will be treated with Therapeutic Exercise;

And a group where will be done Physical Exercise according their preferences.

Pre-intervention, immediate post-intervention, 3 and 6 months assessments will be made. The selection criteria will be: Adult women treated for breast cancer, completed at least 6 months before, with persistent fatigue. All participants must understand and sign freely Informed Consent.

Sample size: 40 women for each group.

Data Analysis: A descriptive analysis of all variables was performed. It establish for all cases a confidence level of 95% (p <0.05). The effectiveness was assessed by comparing the experienced change of the two groups in outcome variables between physical therapy examinations.

ELIGIBILITY:
Inclusion Criteria:

* Women treated for breast cancer, completed at least 6 months before, with persistent fatigue.
* Women who do not present contraindications for physiotherapy and physical exercise (infection, metastasis, loco regional recurrence, cardiopulmonary disorders).
* Women who have read, understood and signed informed consent freely.

Exclusion Criteria:

* Women with cognitive limitations to understand the information provided, instructions for treatment and consent to their participation in the study.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Subjective assessment of perception of fatigue. | 6 months
  FACIT-FatigueScale (total score)

SECONDARY OUTCOMES:
Subjective assessment of perception of dyspnoea | 6 months
  Borg Dyspnoea Test before and after "6-Minutes Walking Test (6MWT)"
Distance in meters | 6 months
  Distance in meters during "6-Minutes Walking Test (6MWT)"
Pain Intensity | 6 months
  Visual analogue scale (VAS).100 mm horizontal with pain descriptors marked "no pain" on the left side or "worst imaginable pain".

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Prieto Go´mez, PhD Student, Principal Investigator — University of Alcalá
Locations (1):
- Teacher care and research in physiotherapy Unit. Department of Physiotherapy. University of Alcala., Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No